CLINICAL TRIAL: NCT03682731
Title: Light Exposure Patterns and Symptoms Among Patients With Erythropoietic Protoporphyria
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ida M. Heerfordt, Principal Investigator, MD, PhD, Bispebjerg Hospital
Other Study IDs: Erythropoietic protoporphyria
Record Dates: First submitted 2018-09-21; First posted 2018-09-25 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Erythropoietic Protoporphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Erythropoietic protoporphyria (EPP) is characterized by development of painful skin symptoms upon exposure to visible light dye to accumulation of the photoactive substance protoporphyrin IX (PpIX) in the skin.This study aimed to quantify the actual light exposure of patients with EPP during everyday life. The investigators further aimed to establish the associations between symptoms and light exposure, use of protective clothes, and erythrocyte PpIX concentration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with erythropoietic protoporphyria
* Informed consent

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with erythropoietic protoporphyria.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Actual light exposure | from April through June 2017
  Actual light exposure of patients with erythropoietic protoporphyria

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen NV

IPD SHARING:
Plan to Share IPD: Undecided